CLINICAL TRIAL: NCT00667706
Title: Prospective Randomized Study of Effects of Laparoscopic Roux-en-Y Gastric Bypass Versus Laparoscopic Sleeve Gastrectomy
Brief Title: Laparoscopic Roux-en-Y Gastric Bypass Versus Laparoscopic Sleeve Gastrectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Carmel Medical Center (Other)
Responsible Party: Andrei Keidar, MD, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBVSSG-HMO-CTIL
Record Dates: First submitted 2008-04-16; First posted 2008-04-28 (Estimated); Last update posted 2008-04-28 (Estimated); Status verified 2008-04

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients who will undergo Laparoscopic Sleeve Gastrectomy
  Interventions: Procedure: laparoscopic operation Sleeve Gastrectomy
- 2 (Active Comparator): Patients who will undergo Laparoscopic Roux-en-Y Gastric Bypass
  Interventions: Procedure: laparoscopic operation Roux-en-Y Gastric bypass

INTERVENTIONS:
Procedure: laparoscopic operation Sleeve Gastrectomy — Laparoscopic Sleeve Gastrectomy will be performed employing a 5-6 trocar technique, and includes gastric resection starting 4-5 cm proximal to the pylorus, using a 38 fr. Bougie and endoscopic stapler with blue and green load.
  Arms: 1
Procedure: laparoscopic operation Roux-en-Y Gastric bypass — Divided LRYGB will employ 5-7 trocars technique, and includes stapled jejunojejunostomy 30-50 cm distal to the Treitz ligament, gastric pouch of 20 cc., and antecolic, antegastric gastrojejunal anastomosis, either two layered hand-sawn, GIA, or EEA-25 -stapled, at surgeons preference. The length of the Roux limb will be 100 centimeters or 150 centimeters in patients with BMI of <50, and >50, respectively.
  Arms: 2

SUMMARY:
The sleeve gastrectomy that has been utilized as a first-stage bariatric procedure to reduce surgical risk in high-risk patients by induction of weight loss is now gaining popularity as a standalone procedure for the treatment of morbid obesity. It appears to be a technically easier and/or faster laparoscopic procedure than Roux-en-Y gastric bypass. It brings good weight loss results, in some studies even comparable to the RYGB and Biliopancreatic Diversion with Duodenal Switch.

The mechanism of action is assumed to be purely restrictive, but some neurohumoral interaction may exist. Almost no data exist on the influence of the sleeve gastrectomy on the medical and general quality of life or resolution of comorbidities.

The rates of the comorbidities resolution 12 to 24 months after sleeve gastrectomy has been reported in the range that seems to be higher than for the purely restrictive procedures.

Our goal is to to compare the surgical and weight loss outcomes between the two procedures, their influence on resolution of common comorbidities and on quality of life change.

150 eligible candidates will be randomized into two groups, one will undergo Laparoscopic Sleeve Gastrectomy, the other will have Laparoscopic Roux-en-Y Gastric Bypass done. Detailed evaluation and preoperative questionnaires will be used to obtain demographic and medical data, and quality of life will be assessed.

General metabolic and nutritional work up will be done, and will be reassessed at different intervals up to 5 years, in order to compare the short and long term results of the two procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with morbid obesity

Exclusion Criteria:

* Pregnancy,
* Previous bariatric operation,
* IBD,
* Previous bowel or stomach surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-04; Primary Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
weight loss | 5 years

SECONDARY OUTCOMES:
short and long term complication rates, length of stay, need for re-operations efficiency of the procedure in inducing weigh loss and resolution of common co-morbidities | 5 years

REFERENCES:
- [Derived] Keidar A, Hershkop KJ, Marko L, Schweiger C, Hecht L, Bartov N, Kedar A, Weiss R. Roux-en-Y gastric bypass vs sleeve gastrectomy for obese patients with type 2 diabetes: a randomised trial. Diabetologia. 2013 Sep;56(9):1914-8. doi: 10.1007/s00125-013-2965-2. Epub 2013 Jun 14. PMID 23765186